CLINICAL TRIAL: NCT05567419
Title: SARS-CoV-2 in Stools Compared to Respiratory Viral Strains, in Patients Hospitalized for COVID-19.
Brief Title: SARS-CoV-2 in Stools Compared to Respiratory Viral Strains.
Acronym: Spread-COVID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Evelyne Schvoerer, Prof. E Schvoerer, Central Hospital, Nancy, France
Other Study IDs: 2022-A00731-42
Record Dates: First submitted 2022-05-24; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stools, respiratory samples, blood samples
  The samples will be studied for viral genome.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Biological assays — PCR and NGS-WGS on stools and respiratory samples

SUMMARY:
The aim of the study is to characterize and to quantify SARS-CoV-2 strains in stools, in comparison with the viral strains in respiratory samples, from patients hospitalized for COVID-19. The methods will be standard ddPCR quantifying SARS-CoV-2 RNA and next generation sequencing-whole genome sequencing. The expected results will allow us to better understand SARS-CoV-2 dynamics and compartmentalization, both in the respiratory tract and in digestive-related tissues, according to the evolution of SARS-CoV-2 variants.

ELIGIBILITY:
Inclusion Criteria:

* Age: men or women of 18 years-old or more
* Clinical signs: hospitalised patient for SARS-CoV-2 infection, nasopharyngeal PCR-confirmed (or any other sample) (in: Infectious diseases department, Intensive care unit), whatever the severity of the clinical form.
* The subject gave his/her informed and writen consent, after complete explanations on the research schedule.
* Compulsory affiliation to a social security scheme.
* Previous medical examination, when a patient is admitted to the hospital, according to good clinical practices.

Exclusion Criteria:

* Subject corresponding to articles L. 1121-5, L. 1121-7 and L1121-8 of the French Public health code:

  * pregnant woman, parturient or breastfeeding woman
  * Minor person
  * Person of full age under guardianship, curatorship, safeguard of justice
* Woman who wants to be pregnant during the study period
* Person in psychiatric care - articles L. 3212-1 and L. 3213-1 who do not fall under the article L. 1121-8 (without consent hospitalisation)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalised patient for SARS-CoV-2 infection, nasopharyngeal PCR-confirmed (or any other sample) in Infectious diseases department and Intensive care unit, whatever the severity of the clinical form.
  n=30
  Sampling dates:
  COVID-19 diagnostics day (d0), day-2, day-4, day-end of hospitalization, day-post hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 dynamics in stools. | 30 monthes
  Evolutive SARS-CoV-2 dynamics in stools compared to respiratory tract: molecular quantification (ddPCR) of SARS-CoV-2 variants genome in stools, compared to the viral quantification in respiratory samples.

SECONDARY OUTCOMES:
SARS-CoV-2 in stools compared to the virus in wastewaters. | 30 monthes
  SARS-CoV-2 in stools compared to wastewaters: molecular quantification (ddPCR) of SARS-CoV-2 variants genome in stools, compared to the viral quantification in wastewater samples.
Modelization of SARS-CoV-2 load in stools and COVID-19 global frequency. | 30 monthes
  SARS-CoV-2 load in stools and COVID-19 global frequency: correlation between SARS-CoV-2 load in stools by ddPCR and COVID-19 incidence in the neighboring global inhabitants population.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne ES Schvoerer, Prof., Principal Investigator — University hospital Nancy, France
Locations (1):
- Schvoerer, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No